CLINICAL TRIAL: NCT02943239
Title: A Randomized, Double-Blind, Placebo-Controlled, Ascending Dose Study to Assess the Safety, Tolerability, and Pharmacodynamic Effects of REGN2477 Alone and in Combination With REGN1033 in Healthy Postmenopausal Women and Healthy Adult Men
Brief Title: Study of Safety, Tolerability, and Pharmacokinetics of REGN2477 Alone and in Combination With REGN1033 in Healthy Postmenopausal Women and Healthy Adult Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: R2477-1033-HV-1621; 2016-002979-95 (EudraCT Number)
Record Dates: First submitted 2016-10-19; First posted 2016-10-24 (Estimated); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- Panel A (Experimental): REGN1033 + REGN2477 (Regimen 1) or placebo
  Interventions: Drug: REGN1033; Drug: REGN2477; Other: Placebo
- Panel B (Experimental): Panel B - REGN1033 + REGN2477 (Regimen 2) or Placebo
  Interventions: Drug: REGN1033; Drug: REGN2477; Other: Placebo
- Panel C (Experimental): Panel C - Patients will receive either REGN1033 + REGN2477 (Regimen 3) or Placebo
  Interventions: Drug: REGN1033; Drug: REGN2477; Other: Placebo
- Panel D (Experimental): Panel D - Patients will receive either REGN1033 + REGN2477 (Regimen 4), REGN1033, REGN2477 (high dose) or Placebo
  Interventions: Drug: REGN1033; Drug: REGN2477; Other: Placebo
- Panel E (Experimental): REGN2477 (Regimen 5) or placebo
  Interventions: Drug: REGN2477; Other: Placebo
- Panel F (Experimental): REGN2477 + REGN1033 (Regimen 6) or placebo
  Interventions: Drug: REGN1033; Drug: REGN2477; Other: Placebo
- Panel G (Experimental): REGN2477 (Regimen 7) or placebo
  Interventions: Drug: REGN2477; Other: Placebo

INTERVENTIONS:
Drug: REGN1033 — REGN1033
  Arms: Panel A; Panel B; Panel C; Panel D; Panel F
Drug: REGN2477 — REGN2477
Other: Placebo — Placebo

SUMMARY:
The primary objective is to assess the safety and tolerability of REGN2477 alone and combined with REGN1033.

The secondary objectives are to:

* Assess the effect of REGN2477 alone, REGN1033 alone, and REGN2477 + REGN1033 in combination on thigh muscle volume
* Assess the effects of REGN2477 alone, REGN1033 alone, and REGN2477 + REGN1033 in combination on total and regional body composition
* Evaluate the Pharmacokinetic (PK) profile of REGN2477 and REGN1033
* Assess immunogenicity of REGN2477 or REGN1033
* Assess REGN2477 or REGN1033 target engagement

ELIGIBILITY:
Key Inclusion Criteria:

* Postmenopausal women age 45 to 70 years and age 35 to 60 years inclusive for men not intending to father children
* BMI between 18 to 32 kg/m2, inclusive
* Willing and able to maintain current diet, supplements and physical activity level throughout the study
* Provides signed informed consent

Key Exclusion Criteria:

* Significant illness or history of significant illness
* Contraindication to MRI
* History of human immunodeficiency virus (HIV); hepatitis B or hepatitis C virus (HCV)
* History of immobilization, major surgical procedure, fracture, or major trauma within 9 months prior to screening
* History of significant gynecological disorders or malignancies; history of breast malignancies (uterine fibroids or dysfunctional uterine bleeding is acceptable)
* Inconsistent vigorous physical activity (on fewer than 5 days per week), such as intermittent weight lifting
* History of hypersensitivity reactions to tetracycline antibiotics (includes doxycycline), vaccines, or biologics
* Use of agents that alter muscle mass that have not been at a stable dose for 3 months prior to screening (includes protein supplements), or use of any weight altering or anabolic steroid drugs (includes drugs for obesity, diuretics, testosterone)
* Participants treated with a biologic therapy or biologic immunotherapy in the previous 12 weeks prior to screening and during the study

Note: Other protocol Inclusion/Exclusion criteria apply.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2016-12-08 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events (TEAEs) | Up to 40 weeks

SECONDARY OUTCOMES:
Percent change in thigh muscle volume as measured by MRI | Up to 28 weeks
Change in thigh muscle volume as measured by MRI | Up to 28 weeks
Percent change in total and regional body composition as measured by Dual X-ray absorptiometry (DXA) | Up to 28 weeks
Change in total body composition as measured by DXA | Up to 28 weeks
Change in regional body composition as measured by DXA | Up to 28 weeks
Pharmacokinetic profile of REGN2477 assessed via measurement of concentrations of REGN2477 in serum over time | Up to 40 weeks
Pharmacokinetic profile of REGN1033 assessed via measurement of concentrations of REGN1033 in serum overtime | Up to 40 weeks
Change in total Activin A levels in blood | Up to 40 weeks
Change in total GDF8 levels in blood | Up to 32 weeks
Presence or absence of antibodies against REGN2477 and REGN1033 | Up to 40 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (2):
- New Zealand (2):
  - Auckland
  - Christchurch

REFERENCES:
- [Derived] Gonzalez Trotter D, Donahue S, Wynne C, Ali S, Parasoglou P, Boyapati A, Mohammadi K, Musser BJ, Meier P, Mastaitis J, Sleeman MW, Glass DJ, Gasparino E, Trejos J, Davis JD, Hirshberg B, Pordy R, Yancopoulos GD, Herman GA. GDF8 and activin A are the key negative regulators of muscle mass in postmenopausal females: a randomized phase I trial. Nat Commun. 2025 May 13;16(1):4376. doi: 10.1038/s41467-025-59380-3. PMID 40360471